CLINICAL TRIAL: NCT05508893
Title: Screening for Coronary Artery Disease USing Primary Evaluation With Coronary Computed Tomography Angiography (CCTA) in Aviation Medicine (SUSPECT)
Brief Title: Screening for Coronary Artery Disease USing Primary Evaluation With Coronary CTA in Aviation Medicine (SUSPECT)
Acronym: SUSPECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding stopped
Sponsor: UMC Utrecht (Other)
Collaborators: Center for Man in Aviation, Royal Netherlands Air Force (Unknown)
Responsible Party: Principal Investigator, Erik Frijters, Principal Investigator, UMC Utrecht
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13-693/D
Record Dates: First submitted 2022-08-09; First posted 2022-08-19 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease (CAD); Coronary Artery Calcification; Occupational Diseases; Aviator's; Disease
MeSH Terms: conditions — Coronary Artery Disease; Occupational Diseases; Disease | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Every participant will perform an exercise test and receive a CTA afterwards
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT Angiography (Other): Coronary CT Angiography will be performed on all individuals
  Interventions: Radiation: CT Angiography
- Exercise stress test (Other): An bicycle exercise stress test will be performed on all individuals
  Interventions: Diagnostic Test: Exercise stress test

INTERVENTIONS:
Radiation: CT Angiography — A CTA will be performed on asymptomatic individuals
  Arms: CT Angiography
Diagnostic Test: Exercise stress test — A routine exercise stress test will be performed on a bicycle
  Arms: Exercise stress test

SUMMARY:
SUSPECT is a prospective, single-center, cohort study of 250 military aircrew at the Center for Man in Aviation, Royal Netherlands Air Force. All asymptomatic aircrew (≥40 years) are asked to undergo a coronary CT scan on a voluntary basis, following the exercise electrocardiograms performed at their routine aeromedical examination. Coronary Artery Calcium score (CACS) and CCTA findings are reported.

ELIGIBILITY:
Inclusion Criteria:

* Military aircrew of the Royal Netherlands Air Force
* ≥ 40 years old
* Required to undergo cardiac screening (per military aviation regulations)

Exclusion Criteria:

* Typical angina
* Prior myocardial infarction
* Prior revascularization therapy (i.e. percutaneous coronary intervention (PCI) and/or coronary artery bypass grafting (CABG))
* Left ventricular ejection fraction <35%
* Does not comprehend study requirements, and/or is unwilling or unable to comply to study procedures
* CT-related contra-indications

  * Allergic to iodine contrast.
  * Renal insufficiency (GFR <60 ml/min/1.73m2, calculated with the Modification of Diet in Renal Disease (MDRD) calculator: http://nephron.org/mdrd_gfr_si.
  * Severe claustrophobia.
  * Uncontrolled irregular heart rhythm or tachycardia unresponsive to beta blockade
  * Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence and severity of CAD in asymptomatic air crew using CCTA as a primary screening tool | 8 Years

SECONDARY OUTCOMES:
Determine the diagnostic accuracy of clinically relevant CAD of the exercise stress test versus CCTA | 8 Years
  Both modalities are used to track down clinically relevant CAD. Clinically relevant CAD is defined as a stenosis of >50%.
Compare the incidence of Major Adverse Cardiac Events (MACE) and all-cause mortality in populations screened between primary and secondary screening after 12 months | 8 Years
Compare the incidence of coronary angiograms and revascularization procedures in the population screened with CTA compared to a historical population using CTA as a secondary screening tool | 8 Years
Establish the additive value of coronary artery calcium score (CACS) in addition to clinical risk scores as a predictor of CAD on CCTA | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Nathoe, PhD, Principal Investigator — UMC Utrecht; Erik Frijters, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Center for Man in Aviation, Soesterberg, Utrecht
  - Utrecht University Medical Center, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frijters E, Nathoe H, Grobben R, Broekhuizen L, Rienks R, Velthuis B. Prevalence and severity of coronary artery disease in asymptomatic military air crew in the Netherlands: a prospective, cross-sectional study (SUSPECT). BMJ Open. 2025 Jun 23;15(6):e100250. doi: 10.1136/bmjopen-2025-100250. PMID 40550709